CLINICAL TRIAL: NCT01366612
Title: PRO#1278: A Phase III Study of Fludarabine and Busulfan Versus Fludarabine, Busulfan and Low Dose Total Body Irradiation in Patients Receiving an Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: PRO#1278: Fludarabine and Busulfan vs. Fludarabine, Busulfan and Total Body Irradiation
Acronym: FLUBUTBI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO#1278: Flu-Bu-TBI
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2022-12-16 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Myeloid Malignancies; Acute Myelogenous Leukemia; Chronic Myelogenous Leukemia; Myeloproliferative Disorders; Myelodysplastic Syndrome
Keywords: Allogeneic Stem Cell Transplant; AML; CML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders; Myelodysplastic Syndromes | interventions — fludarabine; fludarabine phosphate; Busulfan; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): FLUDARABINE AND BUSULFAN
  Interventions: Drug: Fludarabine and Busulfan plus/minus Total Body Irradiation (low dose)
- Group 2 (Experimental): FLUDARABINE, BUSULFAN AND LOW DOSE TOTAL BODY IRRADIATION
  Interventions: Drug: Fludarabine and Busulfan + Low Dose Total Body Irradiation (LD TBI)

INTERVENTIONS:
Drug: Fludarabine and Busulfan plus/minus Total Body Irradiation (low dose) — Fludarabine 40mg/m2 and Busulfan 130mg/m2 on days -6, -5, -4 and -3 of transplant.
  rATG on days -3, -2 and -1
  Other Names: Fludara; Busulfex
  Arms: Group 1
Drug: Fludarabine and Busulfan + Low Dose Total Body Irradiation (LD TBI) — Fludarabine 40mg/m2 and Busulfan 130mg/m2 on days -6, -5, -4 and -3 of transplant.
  rATG on days -3, -2 and -1 TBI 200cGY (as randomized) on day -1
  Other Names: Fludara; Busulfex
  Arms: Group 2

SUMMARY:
This is a single institution study of fludarabine and busulfan versus fludarabine, busulfan and low dose total body irradiation in patients undergoing allogeneic stem cell transplantation. A study population of 80 subjects will be enrolled from The John Theurer Cancer Center at Hackensack University Medical Center. Subjects who are eligible to receive allogeneic hematopoietic stem cell transplantation according to the eligibility criteria will be consented and enrolled. Subjects will be randomly assigned to receive one of 2 conditioning regimen: fludarabine and busulfan, or fludarabine busulfan and low dose total body irradiation (TBI). Subjects will be followed until 1 year post transplantation to assess the relapse rate in each arm and transplant-related toxicity.

The combination of fludarabine and busulfan is the current standard of care for patients with myeloid malignancies (AML, CML and other myeloproliferative disorders, or MDS) undergoing allogeneic transplantation at HUMC. In this study we will be comparing in a randomized fashion the standard regimen to a regimen of fludarabine, busulfan and TBI.

DETAILED DESCRIPTION:
This is a single institution study of fludarabine and busulfan versus fludarabine, busulfan and low dose total body irradiation in patients undergoing allogeneic stem cell transplantation. A study population of 80 subjects will be enrolled from The John Theurer Cancer Center at Hackensack University Medical Center. Subjects who are eligible to receive allogeneic hematopoietic stem cell transplantation according to the eligibility criteria will be consented and enrolled. Subjects will be randomly assigned to receive one of 2 conditioning regimen: fludarabine and busulfan, or fludarabine busulfan and low dose total body irradiation (TBI). Subjects will be followed until 1 year post transplantation to assess the relapse rate in each arm and transplant-related toxicity.

The combination of fludarabine and busulfan is the current standard of care for patients with myeloid malignancies (myelogenous leukemia, chronic myelogenous leukemia, other myeloproliferative disorder, or myelodysplastic syndrome) undergoing allogeneic transplantation at HUMC. In this study we will be comparing in a randomized fashion the standard regimen to a regimen of fludarabine, busulfan and TBI.

Primary Objective The primary objective is to compare the relapse rate at 1 year of patients with myeloid malignancies receiving each regimen.

Secondary Objectives The secondary objective is to compare the toxicity of each regimen

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myelogenous leukemia, chronic myelogenous leukemia, other myeloproliferative disorder, or myelodysplastic syndrome
* Any stage of disease will be considered for transplantation
* Have a suitable related or unrelated donor (Section 3.3)
* Age ≥18 but <70 yrs
* KPS of ≥70%
* Recovery from all hematologic and non-hematology toxicities from previous therapies.

Exclusion Criteria:

* Diagnosis other than acute myelogenous leukemia, myeloproliferative disorder, or myelodysplastic syndrome
* Chemotherapy or radiotherapy within 14 days of initiating treatment in this study with the exception of lenalidomide, decitabine, azacitidine, imatinib mesylate, dasatinib, nilotinib hydrochloride and hydroxyurea
* Prior dose-intense therapy requiring HSC support within 56 days of initiating treatment in this study
* Uncontrolled bacterial, viral, fungal or parasitic infections
* Uncontrolled CNS metastases
* Known amyloid deposition in heart
* Organ dysfunction

  * LVEF <40% or cardiac failure not responsive to therapy
  * FVC, FEV1, or DLCO <50% of predicted and/or receiving supplementary continuous oxygen
  * Evidence of hepatic synthetic dysfunction, or total bilirubin >2x or AST >3x ULN
  * Measured creatinine clearance <20 ml/min
  * Karnofsky score <70%
* Life expectancy limited by another co-morbid illness
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Female subject is pregnant or breast-feeding (women) or unwilling to use acceptable birth control methods (men or women) for twelve months after treatment. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Documented hypersensitivity to fludarabine or melphalan or to bortezomib, boron or mannitol or any components of the formulation
* Patients unable or unwilling to provide consent
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study

Donor Inclusion and Exclusion Criteria

Donor Inclusion Criteria:

HLA 6/6 (HLA-A, B, DrB1) related donor or 7/8 (HLA-A, B, C, DrB1) unrelated donor Related donors will be evaluated in accordance with HUMC standard practice guidelines for the evaluation and management of allogeneic donors Unrelated donors will be identified, evaluated, and managed in accordance with National Marrow Donor Program standards Age ≥18 and <70 yrs KPS of ≥70% Willing to donate bone marrow using standard techniques or peripheral blood HSC by leukapheresis Have adequate veins for apheresis or agree to placement of a central venous catheter (femoral, subclavian) if donating peripheral blood HSC

Donor Exclusion Criteria Identical twin Female donors who are pregnant or breastfeeding Infection with HIV or viral hepatitis (B or C) Known allergy to filgrastim Current serious systemic illness Uncontrolled bacterial, viral, or fungal infection Receiving experimental therapy or investigational agents History of cancer other than treated basal cell cancer of the skin or carcinoma in situ of the cervix. Cancer treated with curative intent >5 yrs before donation will be reviewed on a case-by-case basis by the principal investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-06-16 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Donato, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

REFERENCES:
- [Background] Muller CI, Ruter B, Koeffler HP, Lubbert M. DNA hypermethylation of myeloid cells, a novel therapeutic target in MDS and AML. Curr Pharm Biotechnol. 2006 Oct;7(5):315-21. doi: 10.2174/138920106778521523. PMID 17076647
- [Background] Martin S, Baldock SC, Ghoneim AT, Child JA. Defective neutrophil function and microbicidal mechanisms in the myelodysplastic disorders. J Clin Pathol. 1983 Oct;36(10):1120-8. doi: 10.1136/jcp.36.10.1120. PMID 6311878
- [Background] Martino R, Iacobelli S, Brand R, Jansen T, van Biezen A, Finke J, Bacigalupo A, Beelen D, Reiffers J, Devergie A, Alessandrino E, Mufti GJ, Barge R, Sierra J, Ruutu T, Boogaerts M, Falda M, Jouet JP, Niederwieser D, de Witte T; Myelodysplastic Syndrome subcommittee of the Chronic Leukemia Working Party of the European Blood and Marrow Transplantation Group. Retrospective comparison of reduced-intensity conditioning and conventional high-dose conditioning for allogeneic hematopoietic stem cell transplantation using HLA-identical sibling donors in myelodysplastic syndromes. Blood. 2006 Aug 1;108(3):836-46. doi: 10.1182/blood-2005-11-4503. Epub 2006 Apr 4. PMID 16597592
- [Background] Fukuda T, Hackman RC, Guthrie KA, Sandmaier BM, Boeckh M, Maris MB, Maloney DG, Deeg HJ, Martin PJ, Storb RF, Madtes DK. Risks and outcomes of idiopathic pneumonia syndrome after nonmyeloablative and conventional conditioning regimens for allogeneic hematopoietic stem cell transplantation. Blood. 2003 Oct 15;102(8):2777-85. doi: 10.1182/blood-2003-05-1597. Epub 2003 Jul 10. PMID 12855568
- [Background] Diaconescu R, Flowers CR, Storer B, Sorror ML, Maris MB, Maloney DG, Sandmaier BM, Storb R. Morbidity and mortality with nonmyeloablative compared with myeloablative conditioning before hematopoietic cell transplantation from HLA-matched related donors. Blood. 2004 Sep 1;104(5):1550-8. doi: 10.1182/blood-2004-03-0804. Epub 2004 May 18. PMID 15150081
- [Background] de Lima M, Anagnostopoulos A, Munsell M, Shahjahan M, Ueno N, Ippoliti C, Andersson BS, Gajewski J, Couriel D, Cortes J, Donato M, Neumann J, Champlin R, Giralt S. Nonablative versus reduced-intensity conditioning regimens in the treatment of acute myeloid leukemia and high-risk myelodysplastic syndrome: dose is relevant for long-term disease control after allogeneic hematopoietic stem cell transplantation. Blood. 2004 Aug 1;104(3):865-72. doi: 10.1182/blood-2003-11-3750. Epub 2004 Apr 15. PMID 15090449
- [Background] Andersson BS, de Lima M, Thall PF, Wang X, Couriel D, Korbling M, Roberson S, Giralt S, Pierre B, Russell JA, Shpall EJ, Jones RB, Champlin RE. Once daily i.v. busulfan and fludarabine (i.v. Bu-Flu) compares favorably with i.v. busulfan and cyclophosphamide (i.v. BuCy2) as pretransplant conditioning therapy in AML/MDS. Biol Blood Marrow Transplant. 2008 Jun;14(6):672-84. doi: 10.1016/j.bbmt.2008.03.009. PMID 18489993
- [Background] Bredeson CN, Zhang MJ, Agovi MA, Bacigalupo A, Bahlis NJ, Ballen K, Brown C, Chaudhry MA, Horowitz MM, Kurian S, Quinlan D, Muehlenbien CE, Russell JA, Savoie L, Rizzo JD, Stewart DA. Outcomes following HSCT using fludarabine, busulfan, and thymoglobulin: a matched comparison to allogeneic transplants conditioned with busulfan and cyclophosphamide. Biol Blood Marrow Transplant. 2008 Sep;14(9):993-1003. doi: 10.1016/j.bbmt.2008.06.009. PMID 18721762
- [Background] Russell JA, Savoie ML, Balogh A, Turner AR, Larratt L, Chaudhry MA, Storek J, Bahlis NJ, Brown CB, Quinlan D, Geddes M, Stewart DA. Allogeneic transplantation for adult acute leukemia in first and second remission with a novel regimen incorporating daily intravenous busulfan, fludarabine, 400 CGY total-body irradiation, and thymoglobulin. Biol Blood Marrow Transplant. 2007 Jul;13(7):814-21. doi: 10.1016/j.bbmt.2007.03.003. Epub 2007 Apr 23. PMID 17580259
- [Background] Cox, DR. Regression models and life tables (with discussion). J R Stat Soc B.1972; 34:187-220.
- [Background] Cleveland, WS. Robust locally-weighted regression and smoothing scatterplots. J. Am Stat Assoc. 1979; 74: 829-836.
- [Derived] Suh HC, Rowley SD, Kaur S, Lukasik B, McKiernan P, Boonstra M, Baker M, DiLorenzo M, Skarbnik A, Voss J, Hampson A, DeAgresta B, Boylan B, Nyirenda T, Vesole DH, Donato ML. Prospective, Randomized, Comparative Study of Myeloablative Fludarabine/Busulfan and Fludarabine/Busulfan/Total Body Irradiation Conditioning in Myeloid Diseases. Cancers (Basel). 2025 Mar 28;17(7):1140. doi: 10.3390/cancers17071140. PMID 40227676

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 53 consented, Forty-Seven patients with myeloid diseases were randomized into Flu/Bu4 (25 patients) or Flu/Bu4/TBI (22 patients)
Groups:
- Group 1: FLUDARABINE AND BUSULFAN
  Fludarabine and Busulfan plus/minus Total Body Irradiation (low dose): Fludarabine 40mg/m2 and Busulfan 130mg/m2 on days -6, -5, -4 and -3 of transplant.
  rATG on days -3, -2 and -1
- Group 2: FLUDARABINE, BUSULFAN AND LOW DOSE TOTAL BODY IRRADIATION
  Fludarabine and Busulfan + Low Dose Total Body Irradiation (LD TBI): Fludarabine 40mg/m2 and Busulfan 130mg/m2 on days -6, -5, -4 and -3 of transplant.
  rATG on days -3, -2 and -1 TBI 200cGY (as randomized) on day -1
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 25 | 22
Completed | 25 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 53 consented, Forty-Seven patients with myeloid diseases were randomized into Flu/Bu4 (25 patients) or Flu/Bu4/TBI (22 patients)
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 22 | 47
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 48.4 [23 to 62] | 48.8 [22 to 63] | 48.6 [22 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Relapse Rate at 1 Year of Patients With Myeloid Malignancies Receiving Each Treatment
Time Frame: 1 year
Population: Relapse Rate was analyzed in 34 patients with AML
Measure: Number; unit: Percent
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 18 | 16
Percent | 38.9 | 18.8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 6/25 | 8/22
Serious Adverse Events (participants affected / at risk) | 18/25 | 16/22
Other Adverse Events (participants affected / at risk) | 0/25 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=25) | Group 2 (N=22)
Fever (Investigations) | 1 (1) | 2 (2)
Infection/Reactivation (Infections and infestations) | 5 (5) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
GvHD (Immune system disorders) | 9 (12) | 6 (6)
Relapse/Disease Progression (Investigations) | 7 (7) | 5 (5)
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 1 (1)
BK hemorrhagic cystitis (Infections and infestations) | 0 (0) | 4 (4)
Multi-system failure (Investigations) | 1 (1) | 2 (3)
HUS-TTP (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Vascular disorders) | 0 (0) | 1 (1)
Veno-Occlusive Disease (Vascular disorders) | 0 (0) | 1 (1)
Fall (Investigations) | 0 (0) | 1 (1)
Post-Transplant Lymphoproliferative Disease (Investigations) | 0 (0) | 1 (1)
Colitis and Internal Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sapovirus (Infections and infestations) | 1 (1) | 0 (0)
Limbic Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Acute Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest Pain (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea and Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated LFTs (Investigations) | 0 (0) | 1 (1)
Fever with Nausea and Vomiting (Investigations) | 1 (1) | 0 (0)
Increased Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Left Left Extremity Swelling (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT01366612/Prot_SAP_000.pdf